CLINICAL TRIAL: NCT00399607
Title: Calcium/Vitamin D, Biomarkers & Colon Polyp Prevention
Acronym: PPS4B
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Roberd Bostick, MD, MPH, Professor, Emory University
Other Study IDs: IRB00000357; R01CA114456 (NIH); 0975-2005 (Other: Emory University)
Record Dates: First submitted 2006-11-13; First posted 2006-11-15 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Colorectal Adenomatous Polyps
Keywords: colonic neoplasms; colorectal adenoma; calcium; vitamin D
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Biopsies of normal-appearing rectal mucosa will be collected from participants in an associated parent study.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Aim 1: Participants previously randomized for the parent study will be eligible for a portion of the adjunct biomarker study.
  Interventions: Procedure: Rectal biopsy during colonoscopy
- All aims: Participants entering the parent study will be eligible for all sample collections of the adjunct biomarker study.
  Interventions: Procedure: Rectal biopsy at randomization; Procedure: Rectal biopsy at 1 year; Procedure: Rectal biopsy prior to colonoscopy; Procedure: Biopsies during colonoscopy

INTERVENTIONS:
Procedure: Rectal biopsy during colonoscopy — Biopsies of rectal tissue will be obtained during the 3 or 5 year follow-up colonoscopy. The collection of rectal biopsies involves inserting a tube-about as long and big around as a doctor's examining finger-through the anus into the rectum or lower colon to a depth of about 3-4 inches. At this spot, 4 - 6 tiny pinches of tissue one mm thick (less than 1/16 of an inch) will be taken. The procedure takes less than two minutes, is painless (the only discomfort is like that of having a rectal exam), and is very low risk-about like having blood drawn.
  Groups: Aim 1
Procedure: Rectal biopsy at randomization — Biopsies of rectal tissue will be obtained at the time of randomization. The collection of rectal biopsies involves inserting a tube-about as long and big around as a doctor's examining finger-through the anus into the rectum or lower colon to a depth of about 3-4 inches. At this spot, 4 - 6 tiny pinches of tissue one mm thick (less than 1/16 of an inch) will be taken. The procedure takes less than two minutes, is painless (the only discomfort is like that of having a rectal exam), and is very low risk-about like having blood drawn.
  Groups: All aims
Procedure: Rectal biopsy at 1 year — Biopsies of rectal tissue will be obtained at the time of the one year follow-up visit. The collection of rectal biopsies involves inserting a tube-about as long and big around as a doctor's examining finger-through the anus into the rectum or lower colon to a depth of about 3-4 inches. At this spot, 4 - 6 tiny pinches of tissue one mm thick (less than 1/16 of an inch) will be taken. The procedure takes less than two minutes, is painless (the only discomfort is like that of having a rectal exam), and is very low risk-about like having blood drawn.
  Groups: All aims
Procedure: Rectal biopsy prior to colonoscopy — Biopsies of rectal tissue will be obtained 7-21 days prior to the 3 or 5 year colonoscopy. The collection of rectal biopsies involves inserting a tube-about as long and big around as a doctor's examining finger-through the anus into the rectum or lower colon to a depth of about 3-4 inches. At this spot, 4 - 6 tiny pinches of tissue one mm thick (less than 1/16 of an inch) will be taken. The procedure takes less than two minutes, is painless (the only discomfort is like that of having a rectal exam), and is very low risk-about like having blood drawn.
  Groups: All aims
Procedure: Biopsies during colonoscopy — Biopsies of the rectum, sigmoid colon and ascending colon will be obtained during the 3-5 year follow-up colonoscopy. The colonoscopy involves insertion of a flexible tube through the anus, which is then advanced the full length of the colon. Biopsies (tiny pinches of tissue less than 1/16 of an inch thick) will be taken as the colonoscopy tube is being removed. In total, 12-16 biopsies will be taken from the rectum (or lower colon about 3 - 4 inches up), sigmoid colon and ascending colon.
  Groups: All aims

SUMMARY:
The study team has developed a set of biomarkers of risk for colon cancer; this study tests 1) whether or not calcium and/or vitamin D supplementation can favorably affect these biomarkers in persons who are at higher than average risk for colon cancer (ie, have already undergone the removal of colon growths, called adenomatous polyps, which are known to be precursors to developing colon cancer), and 2) whether effects on the biomarkers predict who will get new colon polyps or not.

DETAILED DESCRIPTION:
This study is an add-on study ('adjunct study') to a clinical trial that is already being conducted (the 'parent study'). Study participants will be composed of persons who are already participating in the parent study, "Vitamin D/Calcium Polyp Prevention Study". In the parent study, a total of 1,964 people nationally are being randomly assigned to four different treatment groups: 1) calcium supplements, 600 mg twice a day; 2) vitamin D supplements, 500 IU twice a day; 3) both the calcium and vitamin D supplements twice a day; and 4) placebo tablets twice a day. The treatment period lasts three to five years at the end of which study participants undergo a follow-up colonoscopy to look for new polyps. The parent study began about a year prior to the start of this adjunct study, thus, there are already some patients in the trial who are receiving their study 'treatments' (i.e., have been 'randomized'), but more patients will be recruited into the parent study.

Depending on whether someone has already been randomized, participants of the parent study will be invited to take part in the adjunct study in one of two ways: 'Aim 1' only, or 'All Aims'. First, patients who have already been randomized will be asked to allow biopsies to be made of their rectal tissue during their 3- or 5-year follow-up colonoscopy (Aim 1). Biopsies, which will be used for our biomarker measurements, are very tiny pieces of tissue that can be examined under the microscope. Second, patients who have not yet been randomized will be invited to participate more fully (All Aims) in the adjunct study. This involves having outpatient rectal biopsies taken immediately after their first phone call, their 1-year follow-up visit, and 7 - 21 days before their 3- or 5-year follow-up colonoscopy. Finally, during their 3- or 5-year colonoscopy, biopsies will be taken from three areas of the colon: the rectum (same area as the outpatient biopsies), the sigmoid colon, and the ascending colon. From all of the biopsies taken from all of the visits and colon sites, biomarker measurements will be of normal proteins that occur in the surface cells lining the colon. Study researchers will then analyze whether calcium and/or vitamin D affect these biomarkers and whether the effects predict who gets new polyps.

ELIGIBILITY:
Currently participating in the parent study. Not open to people not already enrolled in the parent study. This sub-study is for the collection of biopsies only, while the parent study is for calcium and vitamin D to prevent reoccurrence of colon polyps.

Inclusion Criteria for the parent study:

* 45 - 75 years old.
* ≥ 1 histologically-verified neoplastic polyps, ≥ 2 mm in diameter, removed from the large bowel within 4 months of study entry, with entire large bowel examined by colonoscopy and documented free of further polyps.
* Willing to follow the study protocol, as indicated by the subject's informed consent to participate.
* Good general health, with no severely debilitating diseases or active malignancy that might compromise the patient's ability to complete the study.
* Anticipated colonoscopic follow up three years or five years after the qualifying colonoscopy.

Exclusion Criteria for the parent study:

* Invasive carcinoma in any colonic polyp removed.
* Familial colonic polyposis syndromes.
* Ulcerative colitis or Crohn's disease.
* Malabsorption syndrome (e.g., pancreatic insufficiency).
* History of large bowel resection for any reason.
* Diagnosed narcotic or alcohol dependence.
* Elevated serum calcium or creatinine, or supraphysiologic levels of 25(OH) vitamin D at study entry.
* Current use of thiazide diuretic in amount greater than the equivalent of 50 mg of hydrochlorothiazide.
* New York Heart Association Cardiovascular Disease functional class 3 or 4.
* On renal dialysis.
* History of kidney stones, unexplained hematuria, or sarcoidosis in the previous 20 years.
* Any history of hypo- or hyperparathyroidism.
* Unwilling to forgo individual calcium and vitamin D supplementation during the trial.
* Unwilling to forgo daily intake of more than a quart of milk (or equivalent in other dairy products) or daily dietary intake of vitamin D estimated to be greater than 400 IU.
* History of osteoporosis or other medical condition that may require supplemental calcium or vitamin D.
* Current use of bisphosphonates (eg, alendronate [Fosamax], risendronate [Actonel]).
* Current use of calcitonins (eg, Miacalcin).

Additional exclusion criteria for the adjunct biomarker study are:

* Unable to be off aspirin for 7 days.
* History of bleeding disorder or current use of anticoagulant medication.

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in the parent study examining the impact of calcium and vitamin D supplementation on the reoccurrence of colon polyps will be provided the opportunity to also participate in this adjunct biomarker study.
Sampling Method: Non-Probability Sample
Enrollment: 264 (Actual)
Dates: Start 2006-06; Primary Completion 2016-02 (Actual); Study Completion 2016-08 (Actual)

PRIMARY OUTCOMES:
COX-2 Levels | Baseline to end of intervention (up to 5 years)
  Cyclo-oxygenase-2 (COX-2) is an enzyme that is elevated during periods of inflammation. Inflammation and inflammation regulation likely have important roles in colon cancer development. Control of inflammatory response suppresses COX-2.
APC Protein Levels | Baseline to end of intervention (up to 5 years)
  Adenomatous polyposis coli (APC) is a protein encoded by the APC gene and is part of the APC Pathway of colon cancer development. The APC Pathway accounts for familial adenomatosis polyposis (FAP) and approximately 80% of sporadic cancers. The APC protein regulates β-catenin.
β-catenin Levels | Baseline to end of intervention (up to 5 years)
  β-catenin is a protein encoded by the CTNNB1 gene and is part of the APC Pathway of colon cancer development. Overexpression and mutations of β-catenin are associated with multiple cancers, including colorectal cancer. An increase in the ratio of APC to β-catenin is indicative of a decrease of adenoma recurrence.
E-cadherin Levels | Baseline to end of intervention (up to 5 years)
  E-cadherin is a calcium-dependent cell adhesion molecule necessary for colon crypt structure and function. Regulated by β-catenin, E-cadherin is part of the APC Pathway of colon cancer development. An increase in the ratio of APC to E-cadherin is indicative of a decrease of adenoma recurrence.
MLH1 Protein Levels | Baseline to end of intervention (up to 5 years)
  MutL homolog 1 (MLH1) is a protein in the DNA Mismatch Repair (MMR) Pathway. MLH1 protein deficiencies have been found to be related multiple types of cancer, including colorectal cancer. The MMR Pathway accounts for hereditary non-polyosis colon cancer (HNPCC) and approximately 15% of sporadic cancers.
Bax Levels | Baseline to end of intervention (up to 5 years)
  Bax (bcl-2-like protein 4) is a protein that promotes apoptosis of cancer cells and is involved in the DNA Mismatch Repair (MMR) Pathway. Apoptosis is higher in colon neoplasms than in normal colon tissue so a lower expression of bax is indicative of decreased adenoma recurrence.
hTERT Levels | Baseline to end of intervention (up to 5 years)
  hTERT is a catalytic subunit of telomerase. Telomerase is normally present primarily in stem cells and at least some early daughter cells and is expressed in colon and other cancers. A decrease of hTERT is associated in decreased adenoma recurrence.
Bcl-2 Levels | Baseline to end of intervention (up to 5 years)
  B-cell CLL/lymphoma 2 (bcl-2) is a protein encoded by the BCL2 gene which regulates apoptosis. Bcl-2 inhibits apoptosis of abnormal cells. A decrease in the ratio of bax to bcl-2 may be associated with a decrease in adenoma recurrence.
TGFα Levels | Baseline to end of intervention (up to 5 years)
  Transforming growth factor alpha (TGFα), a potent stimulator of colonocyte growth/proliferation, can synergize with c-myc to promote malignant transformation in vitro. A decrease in the ratio of TGFα to TGFβ1 may be associated with a decrease in adenoma recurrence.
TGFβ1 Levels | Baseline to end of intervention (up to 5 years)
  Transforming growth factor beta 1 (TGFβ1), a potent inhibitor of colonocyte growth/proliferation, inhibits c-myc19,26 and induces p21,26 and the growth suppressive activity of TGFβ1 is inhibited by β-catenin (part of the APC Pathway of colon cancer development). A decrease in the ratio of TGFα to TGFβ1 may be associated with a decrease in adenoma recurrence.

CONTACTS AND LOCATIONS:
Overall Officials: Roberd M Bostick, MD, MPH, Principal Investigator — Emory University
Locations (9):
- United States (9):
  - USC/Norris Comprehensice Cancer Center, Los Angeles, California
  - University of Colorado Health Sciences Center, Denver, Colorado
  - Emory University, Atlanta, Georgia
  - University of Iowa Hospitals & Clinic, Iowa City, Iowa
  - University of Minnesota, Minneapolis, Minnesota
  - Dartmouth-Hitchcock Medical Center, Lebanon, New Hampshire
  - University of North Carolina, Chapel Hill, North Carolina
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - University of South Carolina, West Columbia, South Carolina